CLINICAL TRIAL: NCT05041361
Title: HypErthermia as an Additional Treatment for the Biology and Experience of Depression: The HEATBED Study
Brief Title: HypErthermia as an Additional Treatment for the Biology and Experience of Depression
Acronym: HEATBED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEATBED; R34AT011221 (NIH)
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cognitive Behavioral Therapy (CBT) and Whole-Body Hyperthermia (WBH) (Experimental): Participants receive up to 8 weekly (early phase) or 4 bi-weekly (later phase) whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions. Each WBH session (including preparation and cool down) is up to approximately 3.5-4 hours, and each CBT session is approximately 50 minutes.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Device: Whole-Body Hyperthermia (WBH)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician will administer 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
Device: Whole-Body Hyperthermia (WBH) — Whole-body hyperthermia (WBH) will be administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down will last 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH will take place in an infrared sauna dome, and the active heating phase will last until the participants has achieved a core (rectal) temperature of 101.3 F.
  Other Names: Sauna Sessions

SUMMARY:
This single-arm feasibility trial administered up to 8 weekly (early phase) or 4 bi-weekly (later phase) whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions to adults aged 18 years or older with major depressive disorder (MDD).

DETAILED DESCRIPTION:
Major Depressive Disorder afflicts more than 300 million people worldwide and is the leading cause of life years lost to disability. Current treatments have important limitations in efficacy and, in the case of medication, substantial side-effects. There is thus a compelling need for additional effective, well-tolerated treatments. One such potential treatment is whole-body hyperthermia (WBH). The investigators hypothesize that WBH may be particularly effective in combination with cognitive behavioral therapy (CBT), an established treatment for depression. This work holds important promise to improve treatment of depression and advance understanding of the role of integrated mind-body therapies for mood disorders.

This single-arm feasibility trial piloted and optimized procedures for integrating WBH (initially 8 weekly sessions). During the course of this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions were reduced to 4 bi-weekly WBH sessions to improve feasibility.

ELIGIBILITY:
Inclusion criteria:

* Current major depressive episode of at least 4 weeks duration as assessed by the Structured Clinical Interview for DSM-5 (SCID) and a Beck Depression Inventory-II (BDI-II) score greater than or equal to 21 at screening
* Age of at least 18 years old
* Must have smartphone onto which they can download an app from Apple App or Google Play stores
* English speaking
* Ability to lie supine (on back) for 2 hours (required for WBH sessions)
* Must be fully vaccinated against COVID-19

Exclusion criteria:

* Greater than 30 percent reduction in BDI-II score between Screen 1 and Screen 2 (conducted about 1 week after Screen 1)
* Suicide attempt within the prior 12 months and/or severe current suicidal ideation
* Any of the following medical conditions: cardiovascular disease (other than controlled hypertension), seizure disorder, history of cerebrovascular accident (CVA) or other serious neurological condition (e.g. Parkinson's disease, multiple sclerosis, or dementia), current neoplasia, any active enclosed infection (e.g. dental abscess, joint infection), hemophilia or other cause for excessive bleeding (e.g. platelet disorder, or other medical condition that in the opinion of investigators may increase the risk of WBH)
* Comorbid psychiatric conditions or history of comorbid psychiatric conditions that might better explain depressive symptoms, including schizophrenia, schizoaffective disorder, Bipolar Disorder I, Obsessive Compulsive Disorder, Anorexia Nervosa, Bulimia Nervosa, Alcohol Dependence, or Drug Dependence
* Inability to fit into the sauna device
* Known hypersensitivity to hyperthermia and/or infrared exposure
* Breast implants
* Pregnancy, active lactation or intention to become pregnant during the study period

Use of any:

* Medication that might impact thermoregulatory capacity, including: diuretics, barbiturates, beta-blockers, antipsychotic agents, anti-cholinergic agents or chronic use of antihistamines, aspirin (other than low-dose ASA for prophylactic purposes)
* Medication prescribed for the treatment of depression (antidepressant medication; ADM) including but not limited to: selective serotonin reuptake inhibitors [SSRIs], Serotonin and norepinephrine reuptake inhibitors (SNRIs), Monoamine oxidase inhibitors (MAOIs), Tricyclics (TCAs) and atypical antipsychotic and antidepressant medications. Participants must have been free of these medications for at least 4 weeks
* Antibiotics (past 14 days), pain medication (opioids) due to procedure, e.g., dental procedure (past 14 days), emergency contraception pill (past 14 days)
* Medication that in the judgment of the PI would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to WBH
* Recent use (multiple consecutive doses) of: non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, cytokine antagonists
* Greater than 30 percent reduction in Beck Depression Inventory-II (BDI-II) score between Screen 1 and Screen 2
* Has begun new psychotherapy treatment in the prior 6 weeks
* Regular use of any nicotine products, including cigarettes, vapes, chewing tobacco, or other forms of nicotine (if use is not regular, must be willing to refrain for 24 hours before and 24 hours after each WBH session)
* Unwilling to refrain from using marijuana products and alcohol for the 24 hours before and 24 hours after each WBH session
* Unwilling to refrain from sauna use outside of study procedures during study participation, and must not have used a sauna for more than 20 minutes on any single occasion in the 60 days before the screen 2/baseline study visit, and must not have used a sauna in the 30 days before the screen 2/baseline study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco; Frederick M Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janssen CW, Lowry CA, Mehl MR, Allen JJ, Kelly KL, Gartner DE, Medrano A, Begay TK, Rentscher K, White JJ, Fridman A, Roberts LJ, Robbins ML, Hanusch KU, Cole SP, Raison CL. Whole-Body Hyperthermia for the Treatment of Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):789-95. doi: 10.1001/jamapsychiatry.2016.1031. PMID 27172277
- [Background] Hanusch KU, Janssen CH, Billheimer D, Jenkins I, Spurgeon E, Lowry CA, Raison CL. Whole-body hyperthermia for the treatment of major depression: associations with thermoregulatory cooling. Am J Psychiatry. 2013 Jul;170(7):802-4. doi: 10.1176/appi.ajp.2013.12111395. No abstract available. PMID 23820835
- See also: Access to e-screen for interested prospective participants — https://www.sealab.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Midway through this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions (n=6 participants) were reduced to 4 bi-weekly WBH sessions (n=10 participants) to improve feasibility.
Groups:
- Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH): Participants receive up to 8 weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) will be administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasts 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH took place in an infrared sauna dome, and the active heating phase lasts until participants achieved a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician will administer 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
- Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH): Participants receive up to 4 bi-weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) will be administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasts 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH takes place in an infrared sauna dome, and the active heating phase lasts until participants achieved a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician will administer 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH)
Started | 6 | 10
Completed | 5 | 7
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Midway through this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions (n=6 participants) were reduced to 4 bi-weekly WBH sessions (n=10 participants) to improve feasibility.
Groups:
- Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH): Participants receive up to 8 weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) will be administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasts 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH takes place in an infrared sauna dome, and the active heating phase lasts until participants achieve a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician will administer 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
- Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia: Participants receive up to 4 bi-weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) will be administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasts 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH takes place in an infrared sauna dome, and the active heating phase lasts until participants achieve a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician will administer 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (17.3) | 42.4 (9.7) | 41.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 3 | 6 | 9
  African American/Black | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native American | 0 | 0 | 0
  Latino/Hispanic | 0 | 1 | 1
  More Than One Race | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 10 | 16
Beck Depression Inventory-II (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — BDI-II scores range from 0 to 63 with higher scores indicating more severe depression symptoms.
  units on a scale | 27.83 (2.93) | 30.40 (6.64) | 29.44 (5.56)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Planned WBH Sessions Completed
Description: Investigators will average and report the number of completed WBH sessions (4 bi-weekly WBH sessions or 8 weekly WBH sessions offered to participants).
Time Frame: 12 weeks
Population: This feasibility trial piloted and optimized procedures for integrating WBH. The study was planned to be single-arm, but midway through this trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions (n=6 participants) were reduced to 4 bi-weekly WBH sessions (n=10 participants) to improve feasibility; results are here presented separately by number of WBH sessions offered.
Measure: Mean (Standard Deviation); unit: Count of WBH Sessions
Groups:
- Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH): Midway through this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions were reduced to 4 bi-weekly WBH sessions to improve feasibility.
  These results are for participants offered 8 weekly WBH sessions.
  Each WBH session (including preparation and cool down) was up to approximately 3.5-4 hours, and each CBT session is approximately 50 minutes.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician administered 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) was administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasted 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH took place in an infrared sauna dome, and the active heating phase lasted until participants achieved a core (rectal) temperature of 101.3 F.
- Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH): Midway through this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions were reduced to 4 bi-weekly WBH sessions to improve feasibility.
  These results are for participants offered 4 bi-weekly WBH sessions.
  Each WBH session (including preparation and cool down) was up to approximately 3.5-4 hours, and each CBT session is approximately 50 minutes.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician administered 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) was administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasted 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH took place in an infrared sauna dome, and the active heating phase lasted until participants achieved a core (rectal) temperature of 101.3 F.
Arm/Group | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH)
Number analyzed (Participants) | 6 | 10
Count of WBH Sessions | 7.83 (0.41) | 3.20 (1.40)

2. Secondary Outcome: Average Number of Planned Beck Depression Inventory-II (BDI-II) Assessments Completed
Description: Investigators will average and report the number of completed BDI-II assessments (10 planned per participant)
Time Frame: 12 weeks
Population: All participants were offered 8 CBT sessions and administered 10 BDI-II assessments. This feasibility trial piloted and optimized procedures for integrating WBH. The study was planned to be single-arm, but midway through this trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions (n=6 participants) were reduced to 4 bi-weekly WBH sessions (n=10 participants) to improve feasibility; results are here presented separately by number of WBH sessions offered.
Measure: Mean (Standard Deviation); unit: Assessments Completed
Groups:
- Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH): Participants received up to 8 weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) was administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasted 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH took place in an infrared sauna dome, and the active heating phase lasted until participants achieved a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician administered 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
- Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH): Participants received up to 4 bi-weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) was administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasted 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH took place in an infrared sauna dome, and the active heating phase lasted until participants achieved a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician administered 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
Arm/Group | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH)
Number analyzed (Participants) | 6 | 10
Assessments Completed | 9.3 (1.6) | 8.7 (2.6)

3. Secondary Outcome: Change in Beck Depression Inventory-II (BDI-II) From Baseline to 12-week Assessment
Description: Change in BDI-II from baseline assessment to final assessment. BDI-II scores range from 0 to 63 with higher scores indicating more severe depression symptoms.
Time Frame: Baseline and 12 weeks
Population: Midway through this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions (n=6 participants) were reduced to 4 bi-weekly WBH sessions (n=10 participants) to improve feasibility.
  All participants were offered 8 CBT sessions and 10 BDI-II assessments. n=6 offered 8 WBH sessions: n=5 completed the final assessment n=10 offered 4 WBH sessions: n=7 completed the final assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH)
Number analyzed (Participants) | 5 | 7
score on a scale | -16.80 [-27.20 to -6.40] | -15.14 [-25.39 to -4.89]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH): Participants received up to 4 weekly whole-body hyperthermia (WBH) sessions and 8 weekly cognitive behavioral therapy (CBT) sessions.
  Whole-Body Hyperthermia (WBH): Whole-body hyperthermia (WBH) was administered by trained research assistants. Preparation for the WBH, the WBH session, and cool down lasted 3.5-4 hours, with active WBH lasting up to approximately 140 minutes. WBH took place in an infrared sauna dome, and the active heating phase lasted until participants achieved a core (rectal) temperature of 101.3 F.
  Cognitive Behavioral Therapy (CBT): Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician administered 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
Arm/Group | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 5/6 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) and 8 Sessions Whole-Body Hyperthermia (WBH) (N=6) | Cognitive Behavioral Therapy (CBT) and 4 Sessions Whole-Body Hyperthermia (WBH) (N=10)
Lightheadedness (General disorders) | 5 (15) | 3 (4)
Headache (General disorders) | 2 (4) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (4)
Jitteriness (General disorders) | 1 (4) | 0 (0)
Migraine (General disorders) | 1 (2) | 1 (1)
Heat Rash (General disorders) | 1 (2) | 0 (0)
Heart Palpitations (General disorders) | 1 (1) | 1 (1)
Shin Pain (General disorders) | 1 (1) | 0 (0)
Tingling in arms and legs (General disorders) | 1 (1) | 0 (0)
Tinnitus (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose Bowels (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nighttime overheating and body pain (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Midway through this feasibility trial, with oversight and permission from the Sponsor, the 8 weekly WBH sessions (n=6 participants) were reduced to 4 bi-weekly WBH sessions (n=10 participants) to improve feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05041361/Prot_SAP_002.pdf
  • Informed Consent Form (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT05041361/ICF_001.pdf